CLINICAL TRIAL: NCT03968328
Title: The Prognostic Value of the Time From Onset of Fever to Administration of Antibiotics in Neutropenic Fever Patients
Brief Title: Time From Onset of Fever to Administration of Antibiotics in Neutropenic Fever Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0272; NCI-2019-02655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0272 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Febrile Neutropenia; Fever
MeSH Terms: conditions — Febrile Neutropenia; Fever | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview, survey): Patients respond to a survey and participate in an interview with study staff about their fever and when they started feeling unwell.
  Interventions: Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Interview — Take part in interview
Other: Survey Administration — Respond to survey

SUMMARY:
This trial uses an interview and a survey to gather information from cancer patients about the onset of their fever and the administration of antibiotics. Collecting information from patients may help doctors to assess the relationship between time to antibiotic administration and inhospital cause specific death, intensive care unit admission, hospital length of stay, and positive blood cultures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the prognostic value of the length of time between the time onset of fever and first antibiotic administration on cause specific 14 day mortality rate.

SECONDARY OBJECTIVES:

I. To assess the associations of the length of time between the time onset of fever and first antibiotic administration with intensive care unit (ICU) admission, ICU length of stay, length of hospitalization and percentage of patients with positive blood cultures.

OUTLINE:

Patients respond to a survey and participate in an interview with study staff about their fever and when they started feeling unwell.

ELIGIBILITY:
IInclusion criteria:

--> 18 years of age

* Temperature above 38.0 documented
* ANC< 500/mm3

Exclusion Criteria:

--Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the University of Texas MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
14 day cause specific mortality rate | At 14 days
  Will perform univariate logistic regression analysis to assess the effect of time to antibiotic administration on death 14 days post fever onset. Will build multivariate logistic regression model(s) to further assess the effect of time to antibiotic administration on death 14 days post fever onset adjusting for other potential confounders.

SECONDARY OUTCOMES:
Cause specific death | Up to 5 years
Intensive care unit (ICU) admission rate | Up to 5 years
ICU length of stay | Up to 5 years
  Linear regression model will be used to assess the multivariate relationship between time to antibiotic administration, patient demographic and clinical characteristics with ICU length of stay.
Length of hospitalization | Up to 5 years
  Linear regression model will be used to assess the multivariate relationship between time to antibiotic administration, patient demographic and clinical characteristics with length of hospitalization.
Percentage of patients with positive blood cultures | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sai-ching Yeung, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org